CLINICAL TRIAL: NCT00478062
Title: KGEL Vaccine After Initial Therapy of Hodgkin's Lymphoma
Brief Title: Vaccine Therapy in Treating Patients Who Have Received First-Line Therapy for Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J06143 CDR0000544408; P50CA096888 (NIH); P30CA006973 (NIH); JHOC-J06143; JHOC-NA_00007920
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2016-10

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cell vaccine after initial therapy for Hodgkin lymphoma (Experimental): Hodgkin's antigens-GM-CSF-expressing cell vaccine after initial therapy.
  Interventions: Biological: Hodgkin's antigens-GM-CSF-expressing cell vaccine; Procedure: adjuvant therapy

INTERVENTIONS:
Biological: Hodgkin's antigens-GM-CSF-expressing cell vaccine
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines made from a tumor antigen may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and how well vaccine therapy works in treating patients who have received first-line therapy for Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine immunologic responses in patients who have completed first-line therapy for Hodgkin's lymphoma treated with Hodgkin's antigens-GM-CSF-expressing cell vaccine.
* Determine the durability of these immunologic responses in these patients.
* Determine the utility of an Epstein-Barr virus reporter system for monitoring cellular vaccine responses.
* Determine the safety and tolerability of this vaccine in these patients.

OUTLINE: Beginning 4-6 months after last chemotherapy, patients receive Hodgkin's antigens-GM-CSF-expressing cell vaccine on day 1. Treatment repeats every 3 weeks for up to 4 courses.

Immunologic responses are serially monitored along with disease status.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of classic Hodgkin's lymphoma
* Must have completed first-line therapy without evidence of disease progression

PATIENT CHARACTERISTICS:

* HIV negative

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 6 months since prior chemotherapy or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvette L. Kasamon, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cell Vaccine After Initial Therapy for Hodgkin Lymphoma: Hodgkin's antigens-GM-CSF-expressing cell vaccine after initial therapy.
  Hodgkin's antigens-GM-CSF-expressing cell vaccine
  adjuvant therapy
Period: Overall Study
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Immunologic Response
Time Frame: 9 months
Population: The study was closed due to slow accrual, with only one patient enrolled. No data was analyzed for any outcome measures.
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
Number analyzed (Participants) | 0

2. Primary Outcome: Durability of Immunologic Response
Time Frame: 2 years
Population: The study was closed due to slow accrual, with only one patient enrolled. No data was analyzed for any outcome measures.
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
Number analyzed (Participants) | 0

3. Primary Outcome: Utility of Epstein-Barr Virus Reporter System for Monitoring Cellular Vaccine Responses
Time Frame: 2 years
Population: The study was closed due to slow accrual, with only one patient enrolled. No data was analyzed for any outcome measures.
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
Number analyzed (Participants) | 0

4. Primary Outcome: Safety and Tolerability
Time Frame: After administration of last vaccine at 9 weeks
Population: The study was closed due to slow accrual, with only one patient enrolled. No data was analyzed for any outcome measures.
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Cell Vaccine After Initial Therapy for Hodgkin Lymphoma
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes